CLINICAL TRIAL: NCT01388036
Title: A Study in Healthy Subjects to Evaluate Genetic Determinants of the Variability in Hemodynamic Response to Esmolol
Brief Title: Genetic Determinants of Hemodynamic Response to Esmolol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Mordechai Muszkat, MD, Hadassah- Hebrew University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 397-27.05.05
Record Dates: First submitted 2011-07-03; First posted 2011-07-06 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Decrease in Heart Rate Below Baseline Value
Keywords: heart rate
MeSH Terms: interventions — esmolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- esmolol infusion (Experimental): infusion of esmolol during rest and exercise
  Interventions: Drug: esmolol

INTERVENTIONS:
Drug: esmolol — consecutive infusions of esmolol and normal saline (placebo)

SUMMARY:
Beta 1 Adrenergic antagonists (beta blockers) have major role in the treatment of CHF, IHD and hypertension. However, there is large interindividual variability in the response to beta blockers.

The hypothesis underlying this study is that genetic differences between individuals will determine the individual response to esmolol, a betablocker that is administered intravenously. Esmolol will be administered intravenously to healthy volunteers, and the effects on heart rate and blood pressure will be monitored. In addition, we will measure plasma renin activity and plasma levels of norepinephrine.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and female
* able to understand and sign informed consent

Exclusion Criteria:

* consumption of any medication
* bradycardia <50 BPM
* hypersensitivity to beta blockers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate during exercise | 3 hours
  continous measurement of heart rate

SECONDARY OUTCOMES:
change in systolic blood pressure during exercise | 3 hours
  measurement of systolic blood pressure every 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hebrew University Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Muszkat M, Hoofien A, Orlanski-Meyer E, Makhoul H, Porat E, Davidson EM, Blotnick S, Caraco Y. The common Arg389gly ADRB1 polymorphism affects heart rate response to the ultra-short-acting beta(1) adrenergic receptor antagonist esmolol in healthy individuals. Pharmacogenet Genomics. 2013 Jan;23(1):25-8. doi: 10.1097/FPC.0b013e32835afde6. PMID 23114278